CLINICAL TRIAL: NCT06620497
Title: Marginal Bone Loss, Prosthetic and Mucosal Complications of Stress-free Implant Bars and Milled Bars Supporting Mandibular Overdentures. Three-years Randomized Clinical Trial
Brief Title: SFI Bars and Milled Bars Supporting Mandibular Overdentures. Three-year Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Salsabeel A Afifi, PhD, lecturer of oral medicine and periodontology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2492024
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Edentulous Alveolar Ridge in Mandible
Keywords: SFI bar; milled bar; bone loss; mucosal complications; prosthetic complications
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SFI group (Experimental)
  Interventions: Procedure: stress free implant bar
- milled bar group (Active Comparator)
  Interventions: Procedure: milled bar

INTERVENTIONS:
Procedure: stress free implant bar — SFI bar was sectioned and adjusted on the model for more convenience and to save the time of the appointment. The bar (Cendres Metaux, Switzerland) abutments were screwed to the implant analogues.
  Arms: SFI group
Procedure: milled bar — bar abutments were attached to the analogues and scan bodies were threaded into the bar abutments. The cast was scanned using a lab scanner (Ceramill, Amann Girrbach, Germany). The milled bar was selected from the software (Exocad DentalCAD) and designed digitally to connect the implants.
  Arms: milled bar group

SUMMARY:
The aim of this study will be to evaluate the marginal bone loss and prosthetic complications of stress-free implant (SFI) and milled bars used to assist mandibular 4-implant overdentures after 3 years

DETAILED DESCRIPTION:
Eight edentulous participants with insufficient stability of mandibular dentures will receive 4 implants in the mandibular ridge (2 implants in the canine areas and 2 implants in the first molar areas), and then after 3 months, patients will be randomly assigned into 2 groups; 1) group 1: will include 4 participants who will receive milled bar overdentures, and 2) group 2: will include 4 participants who will receive SFI bar overdentures. For both groups, marginal bone loss will be evaluated using the standardized digital periapical films at the time of insertion, 6 months, 1 year, and 3 years after insertion. Prosthetic and mucosal complications will be evaluated after 3 years.

ELIGIBILITY:
Inclusion Criteria:

* mandibular edentulous ridge

Exclusion Criteria:

* severe atrophy in mandibular ridge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
marginal bone loss | time of insertion, 6 months, 1 year and 3 years

SECONDARY OUTCOMES:
prosthetic complications as denture fracture, adjustment of denture margins, acrylic teeth wear/fracture, abutment fracture, abutment screw loosening/fracture, prosthetic screw loosening/fracture, metal housing loosening/wear, clip wear/replacement | 3 years
  include; denture fracture, adjustment of denture margins, acrylic artificial teeth wear or fracture, abutment fracture, abutment screw loosening or fracture, prosthetic screw loosening or fracture, metal housing loosening or wear, plastic clip wear or replacement.
mucosal complications include; mucositis/soreness of mandibular mucosa, ulcer of mandibular mucosa, hyperplasia under the bar | 3 years
  include; mucositis/soreness of mandibular mucosa, ulcer of mandibular mucosa, hyperplasia under the bar

CONTACTS AND LOCATIONS:
Locations (1):
- fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20617218/